CLINICAL TRIAL: NCT03760003
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group, Multiple Dose, Induction Study to Evaluate the Safety, Tolerability and Optimal Dose of ABX464 Compared With Placebo in Patients With Moderate to Severe Ulcerative Colitis Who Have Inadequate Response, Loss of Response, or Intolerance With at Least One of the Following Agents: Immunosuppressant Treatment (i.e. Azathioprine, 6-mercaptopurine, Methotrexate), Tumor Necrosis Factor Alpha [TNF-α] Inhibitors, Vedolizumab, JAK Inhibitors and/or Corticosteroid Treatment
Brief Title: Dose-Ranging Phase 2b Study of ABX464 in Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-103
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
Keywords: ABX464; Refractory patients; Phase 2b; Dose Ranging
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo controlled, parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ABX464 100 mg (Experimental): ABX464 100 mg was administered orally (capsules) once daily for 16 weeks
  Interventions: Drug: ABX464 100 mg
- ABX464 50 mg (Experimental): ABX464 50 mg was administered orally (capsules) once daily for 16 weeks
  Interventions: Drug: ABX464 50 mg
- ABX464 25 mg (Experimental): ABX464 25 mg was administered orally (capsules) once daily for 16 weeks
  Interventions: Drug: ABX464 25 mg
- Matching Placebo (Placebo Comparator): Matching placebo was administered orally (capsules) once daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX464 100 mg — ABX464 100 mg (two capsules of ABX464 50 mg) once daily for 16 weeks
  Other Names: Obefazimod 100 mg
  Arms: ABX464 100 mg
Drug: ABX464 50 mg — ABX464 50 mg (one capsule of ABX464 50 mg + one capsule of placebo) once daily for 16 weeks
  Other Names: Obefazimod 50 mg
  Arms: ABX464 50 mg
Drug: ABX464 25 mg — ABX464 25 mg (one capsule of ABX464 25 mg + one capsule of placebo) once daily for 16 weeks
  Other Names: Obefazimod 25 mg
  Arms: ABX464 25 mg
Drug: Placebo — Two capsules of placebo once daily for 16 weeks
  Other Names: Obefazimod placebo control
  Arms: Matching Placebo

SUMMARY:
Phase 2b study to evaluate the efficacy and the safety of 3 dose-levels of ABX464, administered daily in patients with moderate to severe Ulcerative Colitis.

DETAILED DESCRIPTION:
This phase 2b study will evaluate the efficacy and the safety of 3 dose-levels of ABX464, administered daily in improving Modified Mayo Score (MMS) in patients with moderate to severe Ulcerative Colitis who have inadequate response, loss of response, or intolerance with at least one of the following agents: immunosuppressant treatment (i.e. azathioprine, 6-mercaptopurine, methotrexate), tumor necrosis factor alpha [TNF-α] inhibitors, vedolizumab, JAK inhibitors and/or corticosteroid treatment .

Eligible patients will be randomized into 4 parallel intervention/treatment groups: 100mg q.d of ABX464, 50mg q.d of ABX464, 25mg q.d of ABX464, or matching placebo and will be treated for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 - 75 years;
* Diagnosis of moderate to severe active UC (including ulcerative proctitis if proximal extension of disease occurs beyond 10 cm) confirmed by endoscopy and histology at least 12 Weeks prior to screening visit. Moderate to severe active UC defined by Modified Mayo Score (MMS) of 5 to 9 inclusive (on a scale of 0-9). Moderate to severe active UC should be confirmed at screening visit with a centrally read endoscopy sub-score of at least 2 (on a scale of 0-3);
* Patients having either a documented inadequate response, no response, a loss of response, or an intolerance (defined as the occurrence of at least one Adverse Reaction leading to treatment discontinuation) to either immunosuppressant treatment (i.e., azathioprine, 6-mercaptopurine, methotrexate), tumor necrosis factor [TNF] inhibitors, vedolizumab, JAK inhibitors and/or corticosteroid treatment. Inadequate response, no response, loss of response is defined as:

  i. Active disease or relapse in spite of thiopurines or methotrexate given at an appropriate dose for at least 3 months (i.e. azathioprine 2-2.5 mg/kg/day or mercaptopurine 1-1.5 mg/kg/day in the absence of leukopenia), and/or ii. Active disease despite corticosteroids treatment (prednisolone up to 0.75 mg/kg/day) over a period of 4 Weeks, and/or iii. Active disease or relapse in spite of adequate treatment (as defined in the SmPC) with tumor necrosis factor [TNF] inhibitors or vedolizumab, and/or iv. Active disease or relapse in spite of adequate treatment with JAK inhibitors over a period of at least 6 Weeks.
* Patients receiving oral corticosteroids must have been on a stable dose of prednisone or prednisone equivalent (≤20 mg/day) or on beclomethasone diproprionate (≤5mg/day) or on budesonide MMX (≤9 mg/day) for at least 2 Weeks prior to the screening visit;
* Topical corticosteroids and topical 5-aminosalicylic acid preparations must have been withdrawn at least 2 Weeks prior to the screening visit;
* Patients who are on oral 5-aminosalicylic acid must have been on a stable dose for at least 4 Weeks prior to the screening visit;
* Patients who are receiving immunosuppressants in the form of azathioprine, 6-mercaptopurine, or methotrexate needed to be on a stable dose for at least 4 Weeks prior to screening visit. Patients taking methotrexate also are advised to take folic acid 1 mg/day (or equivalent) supplementation if there is no contraindication;
* Patients on probiotics (e.g., Culturelle® [Lactobacillus GG, i-Health, Inc.], Saccharomyces boulardii) must be on stable doses for at least 2 Weeks prior to the screening visit;
* Patients on antidiarrheals (e.g., loperamide, diphenoxylate with atropine) must be on stable doses for at least 2 Weeks prior to the screening visit;
* Patients who have received tumor necrosis factor [TNF] inhibitors, vedolizumab or other biologics must have discontinued therapy at least 8 Weeks prior to the screening visit due to lack or insufficient efficacy or intolerance;
* Patients previously treated with cyclosporine, tacrolimus or JAK inhibitors must have discontinued therapy at least 4 Weeks prior to the screening visit due to lack or insufficient efficacy or intolerance;
* Patients previously treated with tube feeding, defined formula diets, or parenteral alimentation/nutrition must have discontinued treatment 3 Weeks before the screening visit and must be able to take, orally, appropriate amount of food (calories) and liquids to maintain body weight;
* Patients with surveillance colonoscopy defined as per ECCO guidelines;
* Patients with the following hematological and biochemical laboratory parameters obtained at screening:

  i. Hemoglobin > 9.0 g dL-1; ii. Absolute neutrophil count ≥ 750 mm-3; iii. Platelets ≥ 100,000 mm-3; iv. Total serum creatinine ≤ 1.3 x ULN (upper limit of normal); v. Creatinine clearance > 90 mL min-1 by the Cockcroft-Gault equation within 60 days prior to baseline; vi. Total serum bilirubin < 1.5 x ULN; vii. Alkaline phosphatase, AST (SGOT) and ALT (SGPT) < 2 x ULN;
* Patients are able and willing to comply with study visits and procedures as per protocol;
* Patients should understand, sign and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures are performed;
* Patients should be affiliated to a social security regimen (for French sites only);
* Females and males receiving the study treatment (potentially in combination with immunosuppressant) and their partners must agree to use a highly effective contraceptive method during the study and for 6 months after end of study or early termination. Contraception should be in place at least 2 Weeks prior to study participation. Women must be surgically sterile or if of childbearing potential must use a highly effective contraceptive method. Women of childbearing potential (WOCBP) will enter the study after confirmed menstrual period and a negative pregnancy test. Highly effective methods of contraception include true abstinence, intrauterine device (IUD) or hormonal contraception aiming at inhibition of ovulation, intrauterine hormone releasing system, bilateral tubal ligation, vasectomized partner. True abstinence is defined when this is in line with the preferred and usual lifestyle of the patient. In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is required. This recommendation also applies to WOCBP with an infrequent or irregular menstrual cycle. Female and male patients must not be planning pregnancy during the trial and for 6 months post completion of their participation in the trial. In addition, male participants should use condoms and not donate sperm as long as contraception is required.

Exclusion Criteria:

* Patients with Crohn's Disease (CD) or presence or history of fistula, indeterminate colitis (IC), infectious/ischemic colitis or microscopic colitis (lymphocytic and collagenous colitis);
* History of toxic megacolon, abdominal abscess, symptomatic colonic stricture or stoma; history or imminent colectomy, colonic malignancy;
* History or current evidence of colonic dysplasia or adenomatous colonic polyps. Patient with severe gastrointestinal complications; e.g., short bowel syndromes, recent or planned bowel surgery, Ileostomy and/or colostomy, recent bowel perforation;
* History of more than one episode of herpes zoster or a history (single episode) of disseminated zoster;
* Patients with active infections at screening such as infected abdominal abscess, Clostridium difficile (stool antigen and toxin required), CMV (positive IgM), TB and recent infectious hospitalization;
* Patients previously treated with ABX464;
* Acute, chronic or history of clinically relevant pulmonary, cardiovascular, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable CNS pathology such as seizure disorder, angina or cardiac arrhythmias, active malignancy or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history;
* Acute, chronic or history of immunodeficiency or autoimmune disease;
* History of malignancy excluding patients considered cured (5 years disease free survivors);
* Serious illness requiring systemic treatment and/or hospitalization within 3 Weeks prior to baseline;
* Pregnant or breast-feeding women;
* Illicit drug or alcohol abuse or dependence;
* Patients who received live vaccine 30 days or fewer before first dose of study treatment and/or who's planning to receive such a vaccine during the study duration;
* Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer and during the study;
* Any condition, which in the opinion of the investigator, could compromise the patient's safety or adherence to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Séverine VERMEIRE, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (130):
- United States (4):
  - UCSD Health System, San Diego, California
  - Atlanta Center for Gastroenterology, P.C, Decatur, Georgia
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Ordensklinikum Linz GmbH - Barmherzige Schwestern, Linz
  - AKH - Medizinische Universität Wien, Vienna
- Belarus (5):
  - Gomel Regional Clinical Hospital, Homyel
  - Minsk city diagnostic center, Minsk
  - Regional Clinical Hospital, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
  - Vitebsk regoinal clinical specialized center, Vitebsk
- Belgium (5):
  - AZ Sint-Lucas, Bruges
  - C. H. U. St-Pierre, Brussels
  - UZA, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Canada (6):
  - Brandon Medical Arts Clinic, Brandon
  - South Edmonton Gastroenterology, Edmonton
  - LHSC - Victoria Hospital, London
  - The Ottawa Hospital - General Campus, Ottawa
  - Allen Whey Khye Lim Professional Corporation, Saskatoon
  - Mount Sinai Hospital, Toronto
- Czechia (7):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - MUDr. GREGAR s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Kunčice
  - Nemocnice Na Bulovce, Prague
  - Thomayerova nemocnice, Prague
  - Nemocnice Slany, Slaný
- France (18):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU de Grenoble - Hôpital Nord, Grenoble
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - CHU Lille - Hôpital Claude Huriez, Lille
  - Hôpital Nord - CHU Marseille, Marseille
  - Hopital Saint Eloi, Montpellier
  - CHU Nantes - Hôtel Dieu, Nantes
  - CHU Nice - Hôpital de l'Archet 2, Nice
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg
  - Hopital Rangueil, Toulouse
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (10):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Florence-Nightingale-Krankenhaus-Diakonie Kaiserswerth, Düsseldorf
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Studiengesellschaft BSF Unternehmergesellschaft haftungsbeschraenkt, Halle
  - Universitaetsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Hanover
  - Johanna-Etienne-Krankenhaus, Neuss
  - Tumorzentrum Nordthueringen MVZ GmbH, Nordhausen
  - Dr. Tasso Bieler, Riesa
  - Universitaetsklinikum Ulm, Ulm
- Hungary (7):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem, Debrecen
  - Vasutegeszsegugyi Kft. - Debreceni Egeszsegugyi Kozpont, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
- Italy (10):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - I.R.C.C.S Policlinico San Donato, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello), Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
- Poland (15):
  - Szpital Uniwersytecki nr 2 im.dr J. Biziela, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne Plejady, Krakow
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Wojskowy Szpital Kliniczny w Lublinie, Lublin
  - Trialmed CRS, Piotrkow Trybunalski
  - Centrum Medyczne Grunwald, Poznan
  - KO-MED Centra Kliniczne Pulawy, Puławy
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Centrum Zdrowia MDM, Warsaw
  - Nzoz Vivamed, Warsaw
  - Centrum Zdrowia Tuchow Sp. z o.o., Wierzchosławice
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - LexMedica, Wroclaw
- Serbia (5):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Center Bezanijska Kosa, Belgrade
  - Clinical Center Zvezdara, Belgrade
  - General Hospital Uzice, Užice
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (6):
  - Alian s.r.o., Bardejov
  - Cliniq s.r.o., Bratislava
  - Gastromedic, s.r.o., Nové Zámky
  - Gastro I, s.r.o., Prešov
  - Accout Center s.r.o., Šahy
  - Endomed, s.r.o., Vranov nad Topľou
- Slovenia (3):
  - General Hospital Celje, Celje
  - University Medical Centre Maribor, Maribor
  - General Hospital Murska Sobota, Murska Sobota
- Spain (4):
  - Centro Médico Teknon, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Quironsalud Malaga, Málaga
- Ukraine (17):
  - CNE Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - I.I.Mechnykov Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Central City Clinical Hospital Dept of Theraphy No. 2 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - Communal Non-commercial Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - CI Kherson CCH, Kherson
  - Khmelnytska Regional Hospital, Khmelnytskyi
  - Communal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Regional Clinical Hospital D.Halytskyi Lviv NMU, Lviv
  - Ternopil University Hospital, Ternopil
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - CI City Clinical Hospital #6 Dept of Gastroenterology, Zaporizhzhia
  - CNCE "City Hospital 9" Zaporizhzhia CC, Zaporizhzhia
- United Kingdom (4):
  - Fairfield General Hospital, Bury
  - Guy's Hospital, London
  - University College London Hospitals, London
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 355 patients consented to participate, 254 patients were randomized. A total of 253 patients were treated, 222 patients completed study treatment. 32 patients discontinued and 1 patient was randomized but did not receive study drug. One further patient was excluded from the Full Analysis Set (FAS) due to noncompliance with inclusion/exclusion criteria. A total of 252 patients were included in the FAS (64: ABX464 100mg q.d, 63: ABX464 50mg q.d, 61: ABX464 25mg q.d and 64: placebo).
Pre-assignment Details: Randomization to treatment arms was stratified by previous exposure/non-exposure to biologics and JAK inhibitors treatment use and US/non-US sites.
Groups:
- ABX464 100 mg: ABX464 100 mg was administered orally (two capsules of ABX464 50 mg) once daily for 16 weeks
- ABX464 50 mg: ABX464 50 mg was administered orally (one capsule of ABX464 50 mg + one capsule of placebo) once daily for 16 weeks
- ABX464 25 mg: ABX464 25 mg was administered orally (one capsule of ABX464 25 mg + one capsule of placebo) once daily for 16 weeks
- Matching Placebo: Matching placebo was administered orally (two capsules) once daily for 16 weeks
  Two capsules of placebo once daily for 16 weeks
Period: Overall Study
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Started | 64 | 63 | 63 | 64
Treated | 64 | 63 | 62 | 64
Full Analysis Set | 64 | 63 | 61 | 64
Completed | 54 | 53 | 58 | 57
Not Completed | 10 | 10 | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- ABX464 100 mg: ABX464 100 mg: ABX464 100mg (two capsules of ABX464 50 mg) once daily for 16 weeks
- ABX464 50 mg: ABX464 50 mg: ABX464 50mg (one capsule of ABX464 50 mg + one capsule of placebo) once daily for 16 weeks
- ABX464 25mg: ABX464 25 mg: ABX464 25mg (one capsule of ABX464 25 mg + one capsule of placebo) once daily for 16 weeks
- Matching Placebo: Matching placebo will be administered orally (capsules) once daily for 16 weeks
  Placebo: Two capsules of placebo once daily for 16 weeks
- Total: Total of all reporting groups
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25mg | Matching Placebo | Total
Number analyzed (Participants) | 64 | 63 | 61 | 64 | 252
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 61 | 60 | 56 | 60 | 237
  >=65 years | 3 | 3 | 5 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (12.34) | 40.2 (13.94) | 41.5 (14.16) | 41.1 (14.43) | 41.2 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 36 | 21 | 24 | 104
  Male | 41 | 27 | 40 | 40 | 148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hungary | 5 | 5 | 5 | 7 | 22
  Czechia | 2 | 6 | 4 | 2 | 14
  United States | 0 | 1 | 0 | 1 | 2
  Ukraine | 12 | 7 | 6 | 7 | 32
  Spain | 1 | 0 | 0 | 0 | 1
  Canada | 1 | 1 | 2 | 1 | 5
  Austria | 1 | 1 | 1 | 3 | 6
  Belgium | 4 | 2 | 0 | 2 | 8
  Poland | 16 | 16 | 18 | 20 | 70
  Italy | 5 | 2 | 6 | 7 | 20
  Slovakia | 3 | 7 | 5 | 3 | 18
  Slovenia | 1 | 1 | 1 | 0 | 3
  France | 8 | 8 | 7 | 7 | 30
  Serbia | 0 | 3 | 2 | 0 | 5
  Germany | 5 | 3 | 4 | 4 | 16
Baseline Modified Mayo Score (MMS) [Count of Participants; unit: Participants] — The MMS is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall MMS ranges from 0 to 9 where higher scores represent more severe disease.
  Participants
    Baseline MMS: 4 | 0 | 0 | 0 | 1 | 1
    Baseline MMS: 5 to 6 | 17 | 16 | 17 | 21 | 71
    Baseline MMS: 7 to 9 | 47 | 47 | 44 | 42 | 180

OUTCOME MEASURES:

1. Primary Outcome: Reduction From Baseline in Modified Mayo Score (MMS) at Week 8
Description: Reduction from baseline in Modified Mayo Score (MMS)
  MMS is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall MMS ranges from 0 to 9 where higher scores represent more severe disease.
Time Frame: Week 8
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Groups:
- Matching Placebo: Matching placebo will be administered orally (capsules) and daily for 16 weeks
  Placebo: Two capsules of placebo once daily for 16 weeks orally (Capsules) and daily for 16 weeks
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 58 | 54 | 59 | 60
Score | -2.9 [-3.4 to -2.5] | -3.2 [-3.7 to -2.7] | -3.1 [-3.6 to -2.6] | -1.9 [-2.4 to -1.5]

2. Secondary Outcome: Reduction From Baseline in MMS at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 31 | 30 | 37 | 46
Score
  Overall | -3.6 [-4.3 to -2.9] | -3.2 [-3.9 to -2.5] | -3.3 [-3.9 to -2.7] | -2.4 [-2.9 to -1.8]
  With Previous Biologics or JAK Inhibitors Exposure: number analyzed (Participants) | 21 | 14 | 18 | 23
  With Previous Biologics or JAK Inhibitors Exposure | -3.3 [-4.1 to -2.6] | -3.0 [-3.9 to -2.1] | -2.9 [-3.7 to -2.1] | -1.3 [-2.0 to -0.5]
  Without Previous Biologics or JAK Inhibitors Exposure: number analyzed (Participants) | 10 | 16 | 19 | 23
  Without Previous Biologics or JAK Inhibitors Exposure | -3.6 [-4.8 to -2.3] | -3.4 [-4.4 to -2.5] | -3.7 [-4.6 to -2.8] | -3.4 [-4.2 to -2.6]

3. Secondary Outcome: Number of Participants in Clinical Remission Per MMS at Week 8
Description: Number of participants who achieved clinical remission per Modified Mayo Score at Week 8
  MMS is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall MMS ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical remission is defined as SFS ≤ 1, RBS of 0, and endoscopic subscore ≤ 1 (modified to exclude friability)
Time Frame: Week 8
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 64 | 63 | 61 | 64
Participants | 16 | 11 | 16 | 8

4. Secondary Outcome: Number of Participants in Clinical Remission Per MMS at Week 16
Description: Number of participants who achieved clinical remission per Modified Mayo Score at Week 16
  MMS is a composite score of UC disease activity based on the following 3 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools) to 3 (5 or more stools more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  3. Endoscopic subscore, scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The overall MMS ranges from 0 to 9 where higher scores represent more severe disease.
  Clinical remission is defined as SFS ≤ 1, RBS of 0, and endoscopic subscore ≤ 1 (modified to exclude friability)
Time Frame: Week 16
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 31 | 30 | 37 | 46
Participants | 7 | 6 | 9 | 6

5. Secondary Outcome: Number of Participants With Clinical Response at Week 8
Description: Clinical response is defined as a reduction in MMS of at least 2 points and greater than or equal to 30 percent from baseline with an accompanying decrease in rectal bleeding sub-score of greater than or equal to 1 point or absolute rectal bleeding sub-score of less than or equal to 1 point.
Time Frame: Week 8
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 64 | 63 | 61 | 64
Participants | 32 | 37 | 38 | 22

6. Secondary Outcome: Number of Participants With Clinical Response at Week 16
Description: as for outcome 5
Time Frame: Week 16
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 31 | 30 | 37 | 46
Participants | 19 | 20 | 25 | 20

7. Secondary Outcome: Number of Participants With Endoscopic Improvement at Week 8
Description: Endoscopic improvement is defined as an endoscopic subscore of 0 or 1 (excluding friability)
  Endoscopies were assessed by a blinded central reader and scored according to the following scale:
  0 = Normal or inactive disease;
  1. = Mild disease (erythema, decreased vascular pattern);
  2. = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions);
  3. = Severe disease (spontaneous bleeding, ulceration).
  A higher endoscopic score indicates more severe disease.
Time Frame: Week 8
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 59
Participants | 24 | 21 | 20 | 8

8. Secondary Outcome: Number of Participants With Endoscopic Improvement at Week 16
Description: as for outcome 7
Time Frame: Week 16
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 32 | 31 | 38 | 46
Participants | 11 | 12 | 11 | 9

9. Secondary Outcome: Number of Participants With Mucosal Healing at Week 8
Description: Mucosal healing is defined as endoscopic remission (overall mucosal appearance at endoscopy subscore=0) and histological remission (Geboes score <2.0 based on rectal biopsy).
  The endoscopic subscore ranges from 0 (normal or inactive disease) to 3 (severe disease with spontaneous bleeding, ulceration).
  The Geboes histologic index includes seven histological features (architectural change, chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in epithelium, crypt destruction and erosion or ulcers). The Geboes score has 6 grades, each with 3-5 subgrades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
  A higher score is associated with higher disease activity.
Time Frame: Week 8
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 64 | 63 | 61 | 64
Participants | 0 | 1 | 0 | 2

10. Secondary Outcome: Number of Participants With Mucosal Healing at Week 16
Description: as for outcome 9
Time Frame: Week 16
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 64 | 63 | 61 | 64
Participants | 1 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Reduction of Stool Frequency Relative to Baseline (Day 1)
Description: Participants recorded stool frequency using an electronic subject diary on a daily basis. The stool frequency subscore (SFS) ranges from 0 to 3 according to the following scale:
  Score 0: Normal number of stools Score 1: 1 to 2 stools per day more than normal Score 2: 3 to 4 stools per day more than normal Score 3: 5 or more stools per day more than normal
  Decreasing score indicates improvement.
Time Frame: Day 8, Day 29, Day 57, Day 85, Day 113, and Day 120 (End of Study)
Population: Patients in the category relative to the number of patients in the relevant analysis set and treatment group with data available
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 64 | 63 | 61 | 64
Participants
  Day 8: number analyzed (Participants) | 63 | 61 | 60 | 64
  Day 8 | 18 | 22 | 14 | 12
  Day 29: number analyzed (Participants) | 58 | 57 | 57 | 59
  Day 29 | 34 | 36 | 35 | 26
  Week 8 (Day 57): number analyzed (Participants) | 57 | 52 | 56 | 60
  Week 8 (Day 57) | 39 | 37 | 39 | 37
  Day 85: number analyzed (Participants) | 54 | 51 | 53 | 57
  Day 85 | 41 | 39 | 37 | 30
  Week 16 (Day 113): number analyzed (Participants) | 53 | 52 | 56 | 57
  Week 16 (Day 113) | 44 | 39 | 42 | 38
  End of study (Day 120): number analyzed (Participants) | 6 | 6 | 1 | 2
  End of study (Day 120) | 3 | 4 | 1 | 1

12. Secondary Outcome: Number of Participants With Reduction of Rectal Bleeding Frequency Relative to Baseline
Description: Participants recorded rectal bleeding in an electronic subject diary on a daily basis. Rectal bleeding score (RBS) is taken as the worst subscore of the three most recent scores within 7 days prior to the visit.
  The rectal bleeding subscore ranges from 0 to 3 according to the following scale:
  Score 0: No blood seen Score 1: Streaks of blood with stool less than half the time Score 2: Obvious blood with stool most of the time Score 3: Blood alone passed A lower score represents an improvement in rectal bleeding.
Time Frame: Day 8, Day 29, Day 57, Day 85, Day 113, and Day 120 (End of Study)
Population: Number of participants in the relevant analysis set and treatment group with data available.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 63 | 61 | 60 | 64
Participants
  Day 8 | 25 | 23 | 24 | 16
  Day 29: number analyzed (Participants) | 58 | 57 | 57 | 59
  Day 29 | 44 | 38 | 39 | 24
  Week 8 (Day 57): number analyzed (Participants) | 57 | 53 | 56 | 60
  Week 8 (Day 57) | 48 | 44 | 46 | 33
  Day 85: number analyzed (Participants) | 54 | 51 | 53 | 57
  Day 85 | 47 | 39 | 44 | 35
  Week 16 (Day 113): number analyzed (Participants) | 53 | 52 | 56 | 57
  Week 16 (Day 113) | 50 | 45 | 46 | 37
  End of study (Day 120): number analyzed (Participants) | 6 | 6 | 1 | 2
  End of study (Day 120) | 3 | 4 | 1 | 1

13. Secondary Outcome: Partial Modified Mayo Score Change From Baseline
Description: Partial Modified Mayo Score (pMMS) Change from baseline
  The pMMS is a composite score of UC disease activity based on the following 2 subscores:
  1. Stool frequency subscore (SFS), scored from 0 (normal number of stools per day) to 3 (5 or more stools per day more than normal).
  2. Rectal bleeding subscore (RBS), scored from 0 (no blood seen) to 3 (blood alone passed).
  The overall pMMS score ranges from 0 to 6 with higher scores representing more severe disease.
Time Frame: Day 8, Day 29, Day 57, Day 85, Day 113, and Day 120 (End of Study)
Population: Reduction in least squares mean pMMS for all treatment groups at each visit
Measure: Least Squares Mean (95% Confidence Interval); unit: Score
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 64 | 63 | 61 | 64
Score
  Day 8: number analyzed (Participants) | 63 | 61 | 60 | 64
  Day 8 | -0.7 [-1.0 to -0.3] | -0.8 [-1.1 to -0.4] | -0.7 [-1.0 to -0.4] | -0.4 [-0.7 to -0.1]
  Day 29: number analyzed (Participants) | 58 | 57 | 57 | 59
  Day 29 | -1.8 [-2.1 to -1.5] | -1.8 [-2.2 to -1.5] | -1.8 [-2.1 to -1.4] | -0.9 [-1.3 to -0.6]
  Week 8 (Day 57): number analyzed (Participants) | 58 | 54 | 59 | 60
  Week 8 (Day 57) | -2.2 [-2.6 to -1.9] | -2.2 [-2.5 to -1.9] | -2.3 [-2.6 to -2.0] | -1.6 [-1.9 to -1.3]
  Day 85: number analyzed (Participants) | 54 | 51 | 53 | 57
  Day 85 | -2.4 [-2.8 to -2.1] | -2.3 [-2.6 to -2.0] | -2.3 [-2.7 to -2.0] | -1.6 [-1.9 to -1.3]
  Week 16 (Day 113): number analyzed (Participants) | 53 | 52 | 56 | 57
  Week 16 (Day 113) | -2.8 [-3.1 to -2.4] | -2.4 [-2.8 to -2.1] | -2.6 [-3.0 to -2.3] | -2.0 [-2.3 to -1.7]
  End of Study (Day 120): number analyzed (Participants) | 6 | 6 | 1 | 2
  End of Study (Day 120) | -1.1 [-2.1 to -0.2] | -1.9 [-2.9 to -1.0] | -3.3 [-5.7 to -0.9] | -1.2 [-2.9 to 0.5]

14. Secondary Outcome: Number of Participants With Reduction Relative to Baseline in Fecal Calprotectin at Weeks 8 and 16
Description: Fecal Calprotectin (FC) is a non-invasive surrogate marker of inflammation in the small intestine and levels below 250 ug/g is associated with mucosal healing.
  FC levels were measured using enzyme-linked immunosorbent assay (ELISA) and/or a validated quantitative rapid test. Outcome will be measured based on a reduction in FC relative to baseline values.
Time Frame: Week 8 and Week 16
Population: Number of patients in the relevant analysis set and treatment group, with non-missing values of the parameter
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 44 | 45 | 52 | 52
Participants
  Week 8: number analyzed (Participants) | 44 | 42 | 47 | 52
  Week 8 | 33 | 35 | 33 | 26
  Week 16: number analyzed (Participants) | 44 | 45 | 52 | 43
  Week 16 | 37 | 35 | 37 | 22

15. Secondary Outcome: Number of Participants With Reduction Relative to Baseline in C Reactive Protein at Weeks 8 and 16
Description: CRP is an acute-phase protein which provides an objective criterion of inflammatory activity. CRP has a short half-life (19 hours) and therefore rises early after the onset of inflammation and rapidly decreases after resolution of the inflammation. It is induced by interleukin-6, TNF-alpha and other pro-inflammatory cytokines that are produced within the intestinal lamina propria. Outcome will be measured based on a reduction in CRP relative to baseline values.
Time Frame: Week 8 and Week 16
Population: Number of patients in the relevant analysis set and treatment group, with non-missing values of the parameter
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 58 | 48 | 58 | 58
Participants
  Week 8 (Day 57): number analyzed (Participants) | 58 | 47 | 58 | 58
  Week 8 (Day 57) | 31 | 28 | 39 | 29
  Week 16 (Day 113): number analyzed (Participants) | 54 | 48 | 56 | 57
  Week 16 (Day 113) | 31 | 29 | 37 | 29

16. Secondary Outcome: miRNA-124 Expression (Copy Number) in Whole Blood at Week 8 and Week 16
Description: Absolute quantification (QuantaSoft Pro) of the miR-124 copy number was performed at Week 8 and Week 16 using droplet digital PCR technology (ddPCR) on whole blood samples.
  "0" in the placebo column means "no signal", so BLQ (Below the level of quantification).
Time Frame: Week 8 and Week 16
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Deviation); unit: copies number/cell
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 57 | 50 | 56 | 60
copies number/cell
  Week 8: number analyzed (Participants) | 57 | 47 | 55 | 60
  Week 8 | 13753 (12142) | 8517 (6252) | 4598 (11348) | 28.93 (146.4)
  Week 16: number analyzed (Participants) | 49 | 50 | 56 | 52
  Week 16 | 13268 (11134) | 7723 (7477) | 4154 (5273) | 23.79 (94.69)

17. Secondary Outcome: IL-6 Serum Concentrations
Description: Serum samples from participants who received ABX464 (25, 50 or 100 mg) or placebo were collected during 5 visits (Day 1, Day 8, Day 29, Day 57, and Day 113).
  IL6 was measured using the 8-plex assay on the ELLA Platform (Biotechne). All samples were tested in duplicate at the minimum required dilution.
  Baseline (Day 1) values are calculated as below: x1/arithmetic mean of baseline values x 100, where the arithmetic mean is defined by (x1 + x2+...+xn)/n (summing all baseline values and dividing by the total number of values n)
  The post baseline values are calculated as follow: post-baseline IL-6 values - Day 1 IL-6 values/Day 1 IL-6 values)*100
Time Frame: Day 1
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percentage of IL-6
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 61 | 60 | 64
Percentage of IL-6 | 100 (10.77) | 100 (13.36) | 100 (19.37) | 100 (28.77)

18. Secondary Outcome: Number of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission is defined as an endoscopic subscore of 0.
  Endoscopies were assessed by a blinded central reader and scored according to the following scale:
  0 = Normal or inactive disease;
  1. = Mild disease (erythema, decreased vascular pattern);
  2. = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions);
  3. = Severe disease (spontaneous bleeding, ulceration).
  A higher score represents more severe disease.
Time Frame: Week 8
Population: Number of participants with data for endoscopy relative to the number of patients in the relevant analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 54 | 53 | 58 | 59
Participants | 2 | 5 | 4 | 5

19. Secondary Outcome: Number of Participants With Endoscopic Remission at Week 16
Description: as for outcome 18
Time Frame: Week 16
Population: Number of patients in the category with data available for baseline and the respective visit.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 32 | 31 | 38 | 46
Participants | 1 | 1 | 2 | 3

20. Secondary Outcome: IL-10 Serum Concentrations
Description: Serum samples from patients who received ABX464 (25, 50 or 100 mg) or placebo were collected during 5 visits (Day 1, Day 8, Day 29, Day 57, and Day 113).
  IL10 was measured using the 8-plex assay on the ELLA Platform. All samples were tested in duplicate at the minimum required dilution.
  Baseline (Day 1) values are calculated as below: x1/arithmetic mean of baseline values x 100, where the arithmetic mean is defined by (x1 + x2+...+xn)/n (summing all baseline values and dividing by the total number of values n)
  The post baseline values are calculated as follow: post-baseline IL-10 values - Day 1 IL-10 values/Day 1 IL-10 values)*100
Time Frame: Day 1
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percentage of IL-10
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 61 | 60 | 64
Percentage of IL-10 | 100 (8.982) | 100 (6.989) | 100 (18.98) | 100 (17.54)

21. Secondary Outcome: IL-1B Serum Concentrations
Description: Serum samples from patients who received ABX464 (25, 50, or 100 mg) or placebo were collected during 5 visits (Day 1, Day 8, Day 29, Day 57 and Day 113).
  IL1beta was measured using the 8-plex assay on the ELLA Platform. All samples were tested in duplicate at the minimum required dilution.
  Baseline (Day 1) values are calculated as below: x1/arithmetic mean of baseline values x 100, where the arithmetic mean is defined by (x1 + x2+...+xn)/n (summing all baseline values and dividing by the total number of values n)
  The post baseline values are calculated as follow: post-baseline IL-1B values - Day 1 IL-1B values/Day 1 IL-1B values)*100
Time Frame: Day 1
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percentage of IL-1B
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 62 | 61 | 64
Percentage of IL-1B | 100 (6.514) | 100 (8.988) | 100 (7.043) | 100 (4.87)

22. Secondary Outcome: TNFα Serum Concentrations
Description: Serum samples from patients who received ABX464 (25, 50, or 100 mg) or placebo were collected during 5 visits (Day 1, Day 8, Day 29, Day 57 and Day 113 TNF-alpha was measured using the 8-plex assay on the ELLA Platform. All samples were tested in duplicate at the minimum required dilution.
  Baseline (Day 1) values are calculated as below: x1/arithmetic mean of baseline values x 100, where the arithmetic mean is defined by (x1 + x2+...+xn)/n (summing all baseline values and dividing by the total number of values n)
  The post baseline values are calculated as follow: post-baseline TNFα values - Day 1 TNFα values/Day 1 TNFα values)*100
Time Frame: Day 1
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percentage of TNFα
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 62 | 60 | 64
Percentage of TNFα | 100 (18.79) | 100 (9.313) | 100 (19) | 100 (5.473)

23. Secondary Outcome: Change From Baseline in Infiltrate/Histopathology Using Robarts Histopathology Index (RHI) at Week 8 and Week 16
Description: Infiltrate/Histopathology (Rectal/Sigmoidal Biopsies) using the Robarts Histopathology Index (RHI) Week 8 and Week 16 biopsies will be compared to biopsies at baseline to assess the disease evolution at a tissue level, based on the Robarts Histological Index.
  The score ranges from 0 (no disease activity) to 33 (severe disease activity) is based on evaluation of 4 parameters: chronic inflammatory infiltrate, lamina propria neutrophils and eosinophils, neutrophils in the epithelium and erosion and ulceration.
  A higher score indicates more severe disease.
Time Frame: Week 8 and Week 16
Population: Only samples which were collected have been analyzed. Patients that were evaluated with an endoscopy at week 16 are the subset of patients that did not achieve endoscopic improvement at week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 44 | 44 | 49 | 52
score on a scale
  Week 8 | -7.3 [-9.9 to -4.8] | -5.9 [-8.5 to -3.3] | -7.3 [-9.7 to -4.9] | -3.4 [-5.8 to -1.0]
  Week 16: number analyzed (Participants) | 25 | 18 | 30 | 33
  Week 16 | -7.6 [-11.2 to -4.0] | -5.8 [-10.0 to -1.6] | -8.0 [-11.2 to -4.7] | -2.8 [-5.9 to 0.3]

24. Secondary Outcome: Change From Baseline in Infiltrate/Histopathology - Geboes Score at Week 8 and Week 16
Description: The Geboes score is composed of 6 major grades that assess different aspects of the biopsy findings, with each grade having its own score range:
  1. Structural Changes (Grade 0): Range: 0 (No changes) to 3 (Severe changes)
  2. Chronic Inflammation (Grade 1): Range: 0 (No inflammation) to 3 (Severe inflammation)
  3. Lamina Propria Neutrophils (Grade 2): Range: 0 (None) to 3 (Severe infiltration of neutrophils)
  4. Neutrophils in the Epithelium (Grade 3): Range: 0 (None) to 3 (Severe neutrophil infiltration)
  5. Crypt Destruction (Grade 4): Range: 0 (No destruction) to 3 (Severe crypt destruction)
  6. Erosion and Ulcers (Grade 5): Range: 0 (None) to 3 (Severe erosion/ulceration)
  Subscales are summed across all 6 grades, final total score between 0 and 18 :
  * 0-5: Minimal or no inflammation
  * 6-10: Mild inflammation
  * 11-15: Moderate inflammation
  * 16-18: Severe inflammation or damage A higher score indicates more severe disease
Time Frame: Week 8 and Week 16
Population: Only samples which were collected have been analyzed and included baseline and data for week 8 or week 16. Patients that were evaluated with an endoscopy at week 16 are the subset of patients that did not achieve endoscopic improvement at week 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Score change from baseline
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 44 | 44 | 49 | 52
Score change from baseline
  Week 8 | -4.8 [-6.3 to -3.3] | -3.3 [-4.9 to -1.8] | -4.1 [-5.6 to -2.7] | -1.9 [-3.4 to -0.5]
  Week 16: number analyzed (Participants) | 25 | 18 | 30 | 33
  Week 16 | -4.4 [-6.5 to -2.3] | -3.9 [-6.3 to -1.5] | -4.7 [-6.6 to -2.8] | -1.3 [-3.1 to 0.5]

25. Secondary Outcome: IL-6 Serum Concentrations
Description: as for outcome 17
Time Frame: Day 8, Day 29, Day 57, and Day 113
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 61 | 60 | 64
Percent Change
  Day 8: number analyzed (Participants) | 62 | 60 | 59 | 64
  Day 8 | 166.4 (20.98) | 96.45 (9.034) | 103.6 (8.641) | 132.7 (15.18)
  Day 29: number analyzed (Participants) | 58 | 58 | 59 | 60
  Day 29 | 117 (10.92) | 93.36 (12.19) | 89.31 (8.608) | 128.2 (10.85)
  Week 8 (Day 57): number analyzed (Participants) | 58 | 51 | 60 | 60
  Week 8 (Day 57) | 118.9 (11.3) | 150.6 (47.06) | 89.75 (8.662) | 125.7 (17.11)
  Week 16 (Day 113): number analyzed (Participants) | 52 | 51 | 59 | 57
  Week 16 (Day 113) | 108.3 (14.23) | 170.1 (56.4) | 98.29 (12.03) | 131.8 (16.97)

26. Secondary Outcome: IL-10 Serum Concentrations
Description: as for outcome 20
Time Frame: Day 8, Day 29, Week 8 and Week 16
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 61 | 60 | 64
Percent Change
  Day 8: number analyzed (Participants) | 62 | 60 | 59 | 64
  Day 8 | 100.3 (4.596) | 102.3 (5.827) | 101 (4.288) | 100.1 (3.918)
  Day 29: number analyzed (Participants) | 58 | 57 | 59 | 60
  Day 29 | 98.71 (6.626) | 87.22 (3.638) | 91.40 (4.519) | 102.5 (4.728)
  Week 8 (Day 57): number analyzed (Participants) | 58 | 51 | 60 | 60
  Week 8 (Day 57) | 96.00 (5.590) | 99.30 (7.431) | 89.30 (4.289) | 94.18 (4.886)
  Week 16 (Day 113): number analyzed (Participants) | 52 | 51 | 58 | 57
  Week 16 (Day 113) | 103.9 (7.435) | 92.50 (4.879) | 91.24 (4.911) | 91.85 (5.943)

27. Secondary Outcome: IL-1B Serum Concentrations
Description: as for outcome 21
Time Frame: Day 8, Day 29, Day 57 and Day 113
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 62 | 61 | 64
Percent Change
  Day 8: number analyzed (Participants) | 62 | 60 | 60 | 64
  Day 8 | 102.8 (7.453) | 118.2 (10.44) | 103.7 (5.562) | 111 (5.203)
  Day 29: number analyzed (Participants) | 55 | 57 | 59 | 60
  Day 29 | 115 (9.424) | 101.3 (5.435) | 138 (41.41) | 112.6 (7.052)
  Week 8 (Day 57): number analyzed (Participants) | 56 | 51 | 60 | 60
  Week 8 (Day 57) | 105.3 (5.735) | 100.3 (6.49) | 99 (6.605) | 124.1 (12.24)
  Week 16 (Day 113): number analyzed (Participants) | 52 | 51 | 58 | 57
  Week 16 (Day 113) | 102.4 (6.513) | 137.5 (26.11) | 124.1 (12.24) | 109 (7.042)

28. Secondary Outcome: TNFα Serum Concentrations
Description: as for outcome 22
Time Frame: Day 8, Day 29, Day 57 and Day 113
Population: Only samples which were collected have been analyzed
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | ABX464 100 mg | ABX464 50 mg | ABX464 25 mg | Matching Placebo
Number analyzed (Participants) | 62 | 62 | 60 | 64
Percent Change
  Day 8: number analyzed (Participants) | 62 | 60 | 59 | 64
  Day 8 | 98.8 (3.423) | 96.77 (5.844) | 96.42 (4.552) | 99.7 (2.739)
  Day 29: number analyzed (Participants) | 58 | 57 | 59 | 60
  Day 29 | 99.62 (5.374) | 91.30 (4.676) | 92.64 (4.629) | 110.2 (10.12)
  Week 8 (Day 57): number analyzed (Participants) | 58 | 52 | 60 | 60
  Week 8 (Day 57) | 105.5 (9.675) | 95.55 (4.503) | 97.51 (4.874) | 102.6 (4.873)
  Week 16 (Day 113): number analyzed (Participants) | 52 | 51 | 58 | 57
  Week 16 (Day 113) | 103.7 (7.610) | 108.6 (10.61) | 100.1 (7.194) | 111.4 (7.725)

ADVERSE EVENTS:
Time Frame: TEAEs and SAEs were collected from enrollment to end of study: up to 24 weeks in total, including 4 weeks screening (prior the first dose of study drug), 16 weeks of treatment, and 4 weeks safety follow-up (28 days after last dose of study drug). All-cause mortality was reported from enrollment to end of study: up to 24 weeks in total, including 4 weeks screening (prior the first dose of study drug), 16 weeks of treatment, and 4 weeks safety follow-up (28 days after last dose of study drug).
Description: All AEs and SAEs occurring from the time a patient consents to participate in the study until 4 Weeks after the last dose of study drug.
Groups:
- ABX464, 100mg: ABX464 100mg: ABX464 100mg (two capsules of ABX464 50 mg) once daily for 16 weeks
- ABX464, 50 mg: ABX464 50mg: ABX464 50mg (One capsule of ABX464 50 mg + One capsule of placebo) once daily for 16 weeks
- ABX464, 25mg: ABX464 25mg: ABX464 25mg (One capsule of ABX464 25 mg + One capsule of placebo) once daily for 16 weeks
- Matching Placebo: Matching placebo will be adminstrated orally (Capsules) and daily for 16 weeks
  Placebo: Two capsules of placebo once daily for 16 weeks
Arm/Group | ABX464, 100mg | ABX464, 50 mg | ABX464, 25mg | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63 | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 4/64 | 4/63 | 1/62 | 4/64
Other Adverse Events (participants affected / at risk) | 45/64 | 38/63 | 33/62 | 30/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464, 100mg (N=64) | ABX464, 50 mg (N=63) | ABX464, 25mg (N=62) | Matching Placebo (N=64)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydratation (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464, 100mg (N=64) | ABX464, 50 mg (N=63) | ABX464, 25mg (N=62) | Matching Placebo (N=64)
Headache (Nervous system disorders) | 27 (29) | 19 (21) | 13 (14) | 5 (5)
Burning sensation (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (9) | 4 (5) | 5 (5) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (4) | 3 (4) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dispepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel mouvements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal polip (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotranferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Glutamate Dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio indreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood fibrilogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood fibrilogen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Human chorionic gonadotropin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anal abcsess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes Virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coccydinia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ostheoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyposphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pityriasis Rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis migration (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothiroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mite allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03760003/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03760003/SAP_001.pdf